CLINICAL TRIAL: NCT03758677
Title: A Prospective, Single-center, One-arm Clinical Study of Apatinib Combined With Chemotherapy for Patients Who Progressed After First Line EGFR-TKI Treatment Without T790M Mutation
Brief Title: Apatinib Combined With Chemotherapy for NSCLC Patients Without T790M Mutation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K2018095
Record Dates: First submitted 2018-11-28; First posted 2018-11-29 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — apatinib; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients who progressed after EGFR-TKI without T790M mutation (Experimental): Single arm; Plan to enroll 30 cases; Patients who progressed after EGFR-TKI treatment without T790M mutation
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — 30 patients who progressed after EGFR-TKI treatment without T790M mutation will receive apatinib 250mg qd orally combine with chemotherapy , if the patient has a grade 3/4 adverse reaction during such treatment, apatinib should be reduced to 250mg orally once per two days. Chemotherapeutic agents are limited to platinum-based double drugs(Pemetrexed,Gemcitabine,Docetaxel).
  Other Names: Chemotherapy with platinum-based double drugs(Pemetrexed,Gemcitabine,Docetaxel)

SUMMARY:
At present, with the increasing intensities of the tobacco industry and air pollution in China, the incidence and mortality of lung cancer have become the most important issue that threatens human health.Over the past two decades, the treatment of EGFR+ NSCLC is molecular target therapy (EGFR-TKI). However, only about 30 percent patients with T790M mutation could accept 3rd generation of EGFR-TKI（AZD9291) , most of the patients with progressive disease statuses still stays in the mode of treatment based on radiotherapy and chemotherapy. This is a prospective, single-center, one-arm clinical study designed to evaluate the efficacy and safety of apatinib plus chemotherapy for 30 patients who progressed after EGFR-TKI treatment without T790M mutation. The participants will receive apatinib 250mg qd orally combine with chemotherapy, if the patient has a grade 3/4 adverse reaction during such treatment, it can be reduced to apatinib 250mg orally once per two days. Chemotherapeutic agents are limited to platinum-based double drugs chemotherapy.The primary outcome endpoint was progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

1. male or female patients: 18-75 years old; 2. ECOG performance status score: 0~2 points; 3. Non small cell lung cancer patients who progressed after first line EGFR -TKI treatment without T790M mutation 4.Expected survival period ≥12 weeks; 5.The normal function of major organs, that is, the relevant inspection indicators within the first 14 days of randomness, meet the following requirements:

1. Blood tests:

   1. Hemoglobin ≥ 90 g/L (without transfusion in 14 days);
   2. Neutrophil count ≥ 1.5×109/L;
   3. Platelet count ≥ 100×109/L;
2. Biochemical check:

a .total bilirubin ≤ 1.5 x ULN (upper limit of normal value); b.serum alanine aminotransferase (ALT) or serum aspartate aminotransferase (AST) ≤ 2.5× ULN; if liver metastases, ALT or AST ≤ 5 × ULN; c.Serum creatinine < 1.5 times the upper limit of normal; Endogenous creatinine clearance ≥ 50 ml/min (Cockcroft-Gault formula); 3) Assessment of cardiac Doppler ultrasound: Left ventricular ejection fraction (LVEF) ≥ 50%.

6.Women of childbearing age must have a pregnancy test (serum or urine) within 7 days prior to enrollment, and the result is negative, and they are willing to use appropriate methods of contraception during the trial and within 8 weeks of the last administration of the test drug. For males, consent must be given for contraception or surgical sterilization within 8 weeks of the test period and the last administration of the test drug; 7.Subjects have completely healed after surgery and no bleeding tendency; 8.Good compliance, family members agree to follow the survival follow- up; 9.Sign the informed consent.

Exclusion Criteria:

1. In the past or at the same time suffering from other malignant tumors, 2. Participated in other drug clinical trials within four weeks; 3. Has a variety of factors that affect oral medication (such as inability to swallow, chronic diarrhea, and intestinal obstruction); 4. There is a history of bleeding, and any serious grading within 4 weeks prior to screening has reached 3 degrees or more in CTCAE 4.0; 5. Pre-screening patients with symptomatic central nervous system metastasis or history of central nervous system metastasis; 6. People with high blood pressure who cannot be well controlled by single antihypertensive drugs (systolic blood pressure > 140 mmHg, diastolic blood pressure> 90 mmHg); patients with a history of unstable angina; newly diagnosed angina in the first 3 months before screening or myocardial infarction within 6 months prior to screening; arrhythmia (including QTcF: male ≥450 ms , ≥ 470 ms for females) long-term use of antiarrhythmic drugs and New York Heart Association grade ≥ grade II cardiac insufficiency; 7. Urine prompts urinary protein ≥ ++ and confirmed 24-hour urinary protein quantification> 1.0 g; 8. Combined with anastomotic leakage, duodenal stump fistula, pancreatic fistula or anastomotic stenosis and other serious postoperative complications; 9. Long-term unhealed wounds or incompletely-healed fractures; 10 . Imaging shows that the tumor has invaded an important blood vessel or the investigator judged that the patient's tumor had a high risk of invading vital blood vessels and causing fatal bleeding during treatment; 11. Abnormal coagulation, bleeding tendency (14 days before randomization must meet: in the absence of resistance In the case of coagulants, the INR is within the normal range; Patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin, or the like; International normalized ratio (INR) ≤ 1.5 for prothrombin time Under the premise that small doses of warfarin (1 mg orally, once daily) or low dose aspirin (with daily dose not exceeding 100 mg) are allowed for prophylactic purposes; 12. Incidence of arteriovenous/venous thromboembolism within the first year of screening, such as cerebrovascular accident (including transient ischemic attack), deep venous thrombosis (except for venous thrombosis due to venous catheterization in previous chemotherapy) ) and pulmonary embolism; 13. For female subjects: Surgical sterilization, postmenopausal patients, or agree to use a medically approved contraceptive measure during study treatment and within 6 months of the end of the study treatment period; prior to study enrollment Serum or urine pregnancy tests must be negative within 7 days and must be non-lactating. Male subjects: Should be surgically sterilized, or agree to use a medically-accepted contraceptive treatment during study treatment and within 6 months of the end of the study treatment period; 14. In the past,there was abnormal thyroid function. Even in the case of drug therapy, thyroid function could not be maintained within the normal range.

15. Those who have a history of abuse of psychotropic substances and are unable to get rid of or have mental disorders; 16. Has a history of immunodeficiency, or has other acquired, congenital immunodeficiency disorders, or has a history of organ transplantation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2020-11-20 (Estimated); Study Completion 2021-11-20 (Estimated)

PRIMARY OUTCOMES:
PFS | One to two years
  Progression-free survival

SECONDARY OUTCOMES:
OS | Five years
  Overall survival
AEs | One year
  Adverse events
DCR | One year
  Disease control rate
ORR | One year
  Objective response rate

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China